CLINICAL TRIAL: NCT05647070
Title: Long-term Outcomes of Autologous Transobturator Rectus Fascia Sling for Treatment of Female Stress Urinary Incontinence, Prospective Trial
Brief Title: Long-term Outcomes of Autologous Transobturator Rectus Fascia Sling for Treatment of Female Stress Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, Director, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: autologous transobturator tape
Record Dates: First submitted 2022-11-15; First posted 2022-12-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: A sterile Foley catheter is placed to drain the bladder, following this, injectable normal saline is utilized using 10 cc syringe for hydro-distention of the anterior vaginal wall, and a midline incision is made based on the mid-urethra. Dissection is carried out bilaterally to the obturator Foramen on both sides.
  Through Pfannestiel incision, ~1 cm× ~5 cm rectus fascia strip is isolated from the anterior rectus sheath. Two stay sutures are secured to the corner of the fascial segment on each side. Next, two separate trocar passages are performed on each side using a reusable C-shaped trocar, with care taken to ensure at least a 1 cm tissue bridge in the obturator membrane between the superior and inferior passes. Following this, the stay sutures are tied external to the obturator membrane on both sides, leaving the sling secured and flush with the mid-urethra. Sutures are also placed to secure the sling to the periurethral tissue to prevent rolling or migration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous rectus Fascia TOT (Experimental): A sterile Foley catheter is placed to drain the bladder, following this, injectable normal saline is utilized using 10 cc syringe for hydro-distention of the anterior vaginal wall, and a midline incision is made based on the mid-urethra. Dissection is carried out bilaterally to the obturator Foramen on both sides.
  Through Pfannestiel incision, ~1 cm× ~5 cm rectus fascia strip is isolated from the anterior rectus sheath. Two stay sutures are secured to the corner of the fascial segment on each side. Next, two separate trocar passages are performed on each side using a reusable C-shaped trocar, with care taken to ensure at least a 1 cm tissue bridge in the obturator membrane between the superior and inferior passes. Following this, the stay sutures are tied external to the obturator membrane on both sides, leaving the sling secured and flush with the mid-urethra. Sutures are also placed to secure the sling to the periurethral tissue to prevent rolling or migration
  Interventions: Procedure: Autologous rectus Fascia TOT

INTERVENTIONS:
Procedure: Autologous rectus Fascia TOT — A sterile Foley catheter is placed to drain the bladder, following this, injectable normal saline is utilized using 10 cc syringe for hydro-distention of the anterior vaginal wall, and a midline incision is made based on the mid-urethra. Dissection is carried out bilaterally to the obturator Foramen on both sides.
  Through Pfannestiel incision, ~1 cm× ~5 cm rectus fascia strip is isolated from the anterior rectus sheath. Two stay sutures are secured to the corner of the fascial segment on each side. Next, two separate trocar passages are performed on each side using a reusable C-shaped trocar, with care taken to ensure at least a 1 cm tissue bridge in the obturator membrane between the superior and inferior passes. Following this, the stay sutures are tied external to the obturator membrane on both sides, leaving the sling secured and flush with the mid-urethra. Sutures are also placed to secure the sling to the periurethral tissue to prevent rolling or migration

SUMMARY:
Autologous transobturator sling placement is associated with excellent short-term results and can be performed on an outpatient basis in most cases, so long-term outcomes needs to be verified.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is defined as involuntary passage of urine with rising intra-abdominal pressure. SUI is a common problem affecting 18-26.4% of women.

Over the last two decades, SUI treatment has shifted to a mid-urethral sling (MUS) or a mesh-based bladder neck procedure. Although the surgery was believed to be relatively safe, there has been a steep rise in the number of reported cases of their erosion into the lower urinary tract. Several options outside of synthetic mid-urethral sling placement exist, such as the autologous pubovaginal sling, biologic grafts, or urethral bulking agent injection. Each has its limitations, whether related to morbidity or efficacy.

The autologous slings most commonly used are the fascia lata and the rectus fascia, and they are placed at the urethra-vesical junction through the 'retropubic' approach. In an attempt to present the benefits of a "transobturator" surgical approach and avoiding risks associated with synthetic sling material, Linder and Elliott, 6performed a novel technique for autologous urethral sling placement via a" trans obturator" approach for managing female SUI.

Autologous transobturator sling placement is associated with excellent short-term results and can be performed on an outpatient basis in most cases. Notably, no patients had post-operative voiding dysfunction that necessitated sling release, and there were no major (Clavien III-V) complications.The aim of this study is to report long-term transobturator sling outcomes using autologous rectus fascia for SUI in women.

ELIGIBILITY:
Inclusion Criteria:

* Women with genuine stress urinary incontinence.
* Mixed urinary incontinence with predominant stress element.
* Refractory cases to conservative therapy or patients who are not willing to consider (further) conservative treatment.

Exclusion Criteria:

* Mild Stress urinary incontinence with improvement on conservative therapy or patients refusing surgical treatment.
* Mixed incontinence with predominant Urge urinary incontinence.
* Associated local abnormalities (e.g. cystocele).
* Recent or active urinary tract infection.
* Recent pelvic surgery.
* Neurogenic lower urinary tract dysfunction.
* Previous surgery for stress urinary incontinence.
* Pregnancy
* Less than 12 months post-partum.
* Other gynaecologic pathologies affecting bladder functions ( eg,large fibroids)
* Genito-urinary malignancy.
* Current chemo or radiation therapy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete cure OR improvement of SUI | one year
  Complete cure means no leak on cough stress test and the patient in satisfied on "patient reported outcome".
  Improvement means patient reported leakage only with severe exertion and using a smaller number of pads per day and she feels that she has improved. On examination there was no stress urinary incontinence.
  Failure is considered when patients not fulfilling these criteria

SECONDARY OUTCOMES:
Complications of Autologous TOT | one year
  Measured by clavien-Dindo scoring system
Estimated blood loss | 24 hours
  Blood loss will be estimated by counting up the gauzes and towels used during the procedure [fully soaked gauze = 50 ml blood loss; half-soaked gauze = 30 ml blood loss; fully soaked towel = 150 ml blood loss; half-soaked towel = 75 ml blood loss] (Shorn, 2009).
Operative time | 2 hours
  time consumption from induction of anesthesia till closure of vaginal mucosa

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mohamed Fawzy Salman, Cairo
  - Urology department - Alazhar university, Cairo

IPD SHARING:
Plan to Share IPD: No